CLINICAL TRIAL: NCT00176449
Title: A Comparison of Bupropion SR and Placebo for Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-20763
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine Dependence; Nicotine Use Disorder; Tobacco Dependence; Tobacco-Use Disorder; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion SR (Active Comparator)
  Interventions: Drug: Bupropion SR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Bupropion SR — 150mg twice a day (starting with 150mg once a day for three days)
  Arms: Bupropion SR
Drug: Placebo Oral Tablet — Comparable placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether the adjunctive use of bupropion SR in the context of a psychoeducational program modified for people with schizophrenia might improve the likelihood of successful abstinence in this population. If bupropion SR is effective for reducing cigarette smoking, then it will be important to determine if decreased nicotine intake is associated with a worsening of psychotic, anxiety or depressive symptoms. In addition, it would be important to determine the effect that a reduction in nicotine stimulation would have on patient's cognitive functioning, as nicotinic receptors have been shown to regulate attention and memory function, and it is hypothesized that these functions are normalized by acute nicotine administration in people with schizophrenia

DETAILED DESCRIPTION:
After obtaining consent, patients will enter a two week stabilization phase followed by a 14 week treatment phase. The treatment phase begins with a 9 session group therapy led by clinic nurses trained in the educational model of the American Cancer Association. Subjects will begin the double-blind, randomized, placebo controlled medication phase of treatment following the third group session, which is two weeks prior to the established quit day. Patients will receive either bupropion SR 150mg twice a day (starting with 150mg once a day for three days) or placebo in addition to their usual medication regimen. Patients will be offered the use of nicotine replacement in the form of Nicorette gum from quit day through week 8, the end of the group therapy course. Correct use of the gum will be reviewed in group. Following completion of the group therapy course, patients will continue in their assigned medication group until study completion.

Prior to starting the study, subjects will receive a physical exam and ECG, if they have not had one in the last calendar year. All women will have a pregnancy test, and pregnant women will be excluded from the study. If not already completed, the following Index Assessments will be completed: Demographic forms 1 and 2, SCID, Schedule for the Deficit Syndrome, Patient Psychiatric and Medical History Form. The Fagerstrom Test for Nicotine Dependence, symptom/ functional ratings (BPRS, SANS), Extrapyramidal Rating Scale, body weight, and urinary cotinine levels will be obtained during stabilization and at treatment weeks 2, 4, 8, and 14. The MPRC Side-effect Check List will be obtained week 2 (the start of study medication) and biweekly thereafter throughout the end of the treatment phase. Expired carbon monoxide levels will be measured weekly during the study.

Patients will receive a 60 minute neuropsychological test battery during stabilization and at the end of the study. The test battery will consist of the Rey Auditory Verbal Learning Test, Brief Visuospatial Memory Test, Symbol Digit, Letter Number Sequencing, and Distractibility CPT. Similarly, at stabilization, treatment week 8, and study completion (treatment week 14), subjects will meet with a MIRECC rater to complete a Smoking History (on stabilization only), the Change Assessment Scale, Temptation to Smoke Scale, Decisional Balance Scale, and Smoking Abstinence Self-Efficacy Scale. At these time points they will also have antipsychotic blood levels drawn. Patients will be seen for follow-up assessments at 6 months and one-year. Urine cotinine levels, expired CO levels, and Fagerstrom Test for Nicotine Dependence will be obtained at this time.

A total of fifty subjects will be recruited from the Maryland Psychiatric Research Center, Outpatient Research Program (MPRC ORP), Key Point Southwest Mental Health Center, Revisions, Inc., and The Baltimore, VA. The sample will consist of 50 patients who meet the following inclusion and exclusion criteria:

Inclusion Criteria are:

1. DSM-IV diagnosis of Schizophrenia or schizoaffective disorder
2. Age: 18-64
3. Regular half pack a day smokers
4. Score of at least 4 on the Nicotine Dependency Test

Exclusion Criteria are:

1. Seizure disorders, other Neurologic illnesses, or a family history of seizures
2. A medical condition that could manifest psychiatrically
3. Currently experiencing a depressive episode
4. Active substance abuse
5. Currently receiving bupropion
6. Pregnant women
7. Children (<18 years of age)
8. Two consecutive sodium levels of 130 mmol/L or less

Patients will be paid for their time and any inconvenience they may experience through their participation.

An educational informed consent process will be utilized, and only patients able to give informed and voluntary written consent will be able to participate in the study. Before patients are accepted into the study, they must:

1. give oral and written consent;
2. pass the MPRC evaluation of signed consent test which documents factual understanding of research participation (see Appendix);
3. be aware of alternative treatments, and that alternative clinical care is available;
4. be aware of the right to withdraw, and be aware of the appropriate contact person if they wish to withdraw; and
5. be aware that they may have family members or significant friends involved in the informed consent procedures.

MPRC booklets describing research procedures and clarifying differences between research clinical care and standard clinical care will be made available to potential subjects, referring clinicians, and interested family members. Informed consent forms are previewed by an ad hoc committee to assure MPRC and IRB feedback from the perspectives of family advocates, recipients of care, forensic psychiatry, and service system administration.

Primary outcome measures will be:

1. The Fagerstrom Test for Nicotine Dependence, expired CO level, and urine cotinine will be used to determine if bupropion SR, when used as an adjunct to antipsychotic medication, is superior to placebo for helping patients with schizophrenia improve their chances of smoking cessation.
2. Neuropsychological testing will be used to determine the effects of smoking cessation on patient's attention and memory function.

Secondary outcome measures will be:

1. BPRS, SANS, EPRS, and body weight will be used to determine the effects of bupropion SR and smoking cessation on patients' positive and negative symptoms, level of functioning, and physical health.
2. To determine whether responses to the Smoking Consequences Questionnaire, Change Assessment Scale, Temptation to Smoke Scale, Decisional Balance Scale, and Smoking Abstinence Self-Efficacy Scale correlate with successful smoking cessation.

In a preliminary study, we were able to detect a 44% reduction in expired CO with bupropion treatment. This represents a change in 1.2 SDs, a large effect size. In order to detect the same effect in the proposed double-blind study, with two-sided tests at alpha=.05 and power of 0.80, we would need 10 subjects in each treatment group. Since open labeled study designs may inflate observed effects, we have decide to include 20 subjects in each group. The primary analytic approach will use repeated measures ANCOVA, with adjustment for baseline expired CO level, with treatment assignment as the between group factor and expired CO level as the repeated measure. Since both groups will receive group therapy, the value at the end of the first week of group (before starting bupropion or placebo) will be used as the baseline for comparing patients on bupropion versus placebo. A similar approach will be used to analyze the symptom and neurocognitive measures.

The major risks of the study are the stress of and symptoms associated with nicotine withdrawal. Depressed mood, insomnia, irritability, anger, anxiety, difficulty concentrating, restlessness, decreased heart rate, and increased appetite are all common. Risks associated with the use of bupropion SR include allergic reactions (most commonly skin rashes and itching), dry mouth, insomnia, dizziness, tremor, and headaches. Of these, dry mouth and insomnia are most common. The risk of seizure, when using sustained -release bupropion in the dose range used in this study, is 0.1%, a rate similar to that of other antidepressants. Because bupropion is a weak dopamine agonist, it is possible that subjects may experience a worsening of psychosis. However, work at the MPRC ORP and other places with similar dopamine agonists showed there was no worsening in baseline psychotic symptoms, when patients remained on antipsychotics. There are studies to support the safety of combining antipsychotic medications with selective serotonin reuptake inhibitors and bupropion. However, there is always the potential for unforeseen drug interactions, with the addition of bupropion to existing medication regimens.

Use of Nicorette gum has been associated with sore throat or mouth, hiccups, tired jaws, nausea or other gastrointestinal symptoms, and rarely mouth ulcers. Nicotine intoxication from overuse of the gum is unlikely, as it is released slowly from the gastrointestinal tract and undergoes extensive presystemic metabolism.

The neuropsychological tests are associated with minimal risks. Some subjects may find the testing stressful or boring. The likelihood of this occurring is unlikely. However, frequent breaks in the testing will be allowed to insure that the subject does not become overwhelmed.

To protect privacy and confidentiality, the patient's welfare will be safeguarded by responsible, systematically controlled procedures in the collection of information for both research and clinical purposes. Recorded information for research purposes will be identified by code number rather than by name. Information gathered will be kept in a research chart maintained in a locked file cabinet. Published or presented material related to the project will not be traceable to specific individuals.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria are:

  1. DSM-IV diagnosis of Schizophrenia or schizoaffective disorder
  2. Age: 18-64
  3. Regular half pack a day smokers
  4. Score of at least 4 on the Nicotine Dependency Test

     Exclusion Criteria:

     Exclusion Criteria are:

  <!-- -->

  1. Seizure disorders, other Neurologic illnesses, or a family history of seizures
  2. A medical condition that could manifest psychiatrically
  3. Currently experiencing a depressive episode
  4. Active substance abuse
  5. Currently receiving bupropion
  6. Pregnant women
  7. Children (<18 years of age)
  8. Two consecutive sodium levels of 130 mmol/L or less

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2001-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The Fagerstrom Test for Nicotine Dependence, expired CO level, and urine cotinine will be used to determine if bupropion SR, when used as an adjunct to antipsychotic medication, is superior to placebo for helping patients with schizophrenia improve their | Expired CO weekly, Fagerstrom baseline and end of study, Urine cotinine baseline, week 2 and week 8
Neuropsychological testing will be used to determine the effects of smoking cessation on patient's attention and memory function. | Beginning and end of study

SECONDARY OUTCOMES:
BPRS, SANS, EPRS, and body weight will be used to determine the effects of bupropion SR and smoking cessation on patients' positive and negative symptoms, level of functioning, and physical health. | Baseline, week 2, 4, 8, and 14
To determine whether responses to the Smoking Consequences Questionnaire, Change Assessment Scale, Temptation to Smoke Scale, Decisional Balance Scale, and Smoking Abstinence Self-Efficacy Scale correlate with successful smoking cessation. | Beginning and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Elaine E Weiner, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric REsearch Center, Catonsville, Maryland, United States

REFERENCES:
- [Result] Weiner E, Ball MP, Summerfelt A, Gold J, Buchanan RW. Effects of sustained-release bupropion and supportive group therapy on cigarette consumption in patients with schizophrenia. Am J Psychiatry. 2001 Apr;158(4):635-7. doi: 10.1176/appi.ajp.158.4.635. PMID 11282701
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Agarwal SM, Stogios N, Ahsan ZA, Lockwood JT, Duncan MJ, Takeuchi H, Cohn T, Taylor VH, Remington G, Faulkner GEJ, Hahn M. Pharmacological interventions for prevention of weight gain in people with schizophrenia. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013337. doi: 10.1002/14651858.CD013337.pub2. PMID 36190739
- [Derived] Weiner E, Ball MP, Buchholz AS, Gold JM, Evins AE, McMahon RP, Buchanan RW. Bupropion sustained release added to group support for smoking cessation in schizophrenia: a new randomized trial and a meta-analysis. J Clin Psychiatry. 2012 Jan;73(1):95-102. doi: 10.4088/JCP.10m06143gre. Epub 2011 Apr 5. PMID 21535998